CLINICAL TRIAL: NCT05496530
Title: One Year Results for Suprachoroidal Triamcinolone Acetonide Injection in Various Retinal Diseases
Brief Title: Custom Needle Preparation for Suprachoroidal Steroid Injection (One Year Results)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelshafy, Lecturer of Ophthalmology, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rc-11-22
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Diabetic Macular Edema; Vogt Koyanagi Harada Disease; Retinal Vein Occlusion
MeSH Terms: conditions — Uveomeningoencephalitic Syndrome; Retinal Vein Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diabetic macular edema (Active Comparator): Cases with diabetic macular edema with central macular thickness more than 300 microns measured by optical coherence tomography.
  Interventions: Drug: Suprachoroidal triamcinolone acetonide injection
- Vogt-koyanagi harada (Active Comparator): Cases with vogt-koyanagi harada and complicated with exudative retinal detachment confirmed by optical coherence tomography.
  Interventions: Drug: Suprachoroidal triamcinolone acetonide injection
- Retinal vein occlusion (Active Comparator): Cases with retinal vein occlusion and complicated with macular edema confirmed by optical coherence tomography.
  Interventions: Drug: Suprachoroidal triamcinolone acetonide injection

INTERVENTIONS:
Drug: Suprachoroidal triamcinolone acetonide injection — Pars plana suprachoroidal injection of 4mg//0.1ml triamcinolone acetonide.

SUMMARY:
Suprachoroidal drug delivery is a recent route for managing various ocular conditions. Safety and long term results are still under investigations.

DETAILED DESCRIPTION:
In this study, we aim to analyze the long term results of suprachoroidal injection in treating various retinal diseases to focus on its efficacy, safety and long term ocular effects as ocular hypertension, cataract progression and macular edema resolution.

ELIGIBILITY:
Inclusion Criteria:

* cases with central macular thickness more than 250 microns measured by optical coherence tomography due to one of the following conditions:
* Diabetic macular edema
* Vogt-koyanagi Harada disease
* Retinal vein occlusion.

Exclusion Criteria:

* other causes of increased macular thickness as age related macular degeneration and myopic choroidal new vascularization.
* Cases with confirmed diagnosis of glaucoma.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-10 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | Baseline and up to one year after injection.
  Changes noted in vision after injection measured 8n logMar units by snellen chart.

SECONDARY OUTCOMES:
Central macular thickness | Baseline and up to one year after injection.
  Changes noted in central macular thickness after injection measured by optical coherence tomography in microns.

OTHER OUTCOMES:
Intraocular pressure | Baseline and up to one year after injection.
  Changes noted in intraocular pressure after injection measured by applanation tonometry in millimeter mercury.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Tabl, Principal Investigator — Benha University
Locations (1):
- Ahmed Abdelshafy Tabl, Banhā, Benha, Egypt